CLINICAL TRIAL: NCT03731611
Title: Impact of Umbilical Cord Milking in Preterm Neonates With Placental Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Professor of pediatrics/Neonatology, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS/17.07.44
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Placental Insufficiency; Preterm Infant
Keywords: Umbilical cord milking
MeSH Terms: conditions — Placental Insufficiency; Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): umbilical cord milking will be done for preterm infants <34 gestational age without placental insufficiency
  Interventions: Procedure: Umbilical Cord Milking
- Group B (Active Comparator): umbilical cord milking will be done for preterm infant <34 gestational age with placental insufficiency
  Interventions: Procedure: Umbilical Cord Milking
- Group C (No Intervention): Immediate cord clamping for preterm infants <34 gestational age with placental insufficiency

INTERVENTIONS:
Procedure: Umbilical Cord Milking — Umbilical cord milking (UCM) is typically performed by placing the infant below the level of the placenta. The cord is held at 20-25 cm distance from the baby and milked vigorously towards the umbilicus for 3 times at a speed of 10 cm/sec. After completion, the cord is clamped, and the neonate is handed to the resuscitation team.
  Arms: Group A; Group B

SUMMARY:
To investigate the effect of umbilical cord milking (UCM) on peripheral hematologic parameters including hematopoietic progenitor cells in premature infants ≤ 34 weeks gestational age with placental insufficiency. We hypothesize that UCM would enhance peripheral CD34 concentration, hemoglobin and reduce prematurity complications like NEC and IVH in preterm infant ≤ 34 week gestational age with placental insufficiency.

DETAILED DESCRIPTION:
A pilot prospective randomized controlled study will be conducted among 3 groups, all of them are preterm less than 34 weeks gestational age, in the first group umbilical cord milking will be done for preterm infant with placental insufficiency. Two control groups are present, in the first one umbilical cord milking will be done for preterm infants without placental insufficiency (Insufficiency vs. no insufficiency), another group of immediate cord clamping for preterm infants with placental insufficiency will be added (milking vs. no milking), 30 cases will be recruited in each group.

Umbilical cord milking (UCM) is typically performed by placing the infant below the level of the placenta. The cord is held at 20-25 cm distance from the baby and milked vigorously towards the umbilicus for 3 times at a speed of 10 cm/sec. After completion, the cord is clamped, and the neonate is handed to the resuscitation team.

One milliliter of fetal blood will be taken from peripheral venous blood in the first 30 min of life and CD34 will be assessed by flow cytometry. Secondary outcomes will be documented during NICU stay that include admission CBC, peak bilirubin concentrations, CBC after 2 months, neonatal morbidity such as sepsis, bronchopulmonary dysplasia, necrotizing enterocolitis, retinopathy of prematurity and polycythemia, therapeutic interventions such as need for inotropes, nasal CPAP, mechanical ventilation and phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates < 34 weeks gestational age

Exclusion Criteria:

* Vaginal bleeding due to placental abruption or tears
* Multiple pregnancies
* Suspected major fetal anomalies
* Suspected chromosomal aberration
* Maternal drug abuse
* Hydrops fetalis
* preterm who needed major resuscitative measures

Min Age: 0 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Peripheral venous CD34 at admission | first 24 hours of infants' life
  One milliliter of fetal blood will be taken from peripheral venous blood in the first 30 min of life and CD34 will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Admission hemoglobin | first 24 hours of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood in the first 24 hours of life.
Hemoglobin at 2 months | 2 months after umbilical cord milking
  One milliliter of neonatal blood will be taken from peripheral venous blood at 2 months of life.
Admission platelets | first 24 hours of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood in the first 24 hours of life.
Admission WBCs | first 24 hours of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood in the first 24 hours of life.
Phototherapy requirements | first 28 days of life
  Need to start phototherapy for hyperbilirubinemia
Polycythemia | first 28 days of life
  arterial Hematocrit value more than 70%
Culture proven sepsis | first 28 days of life
  Sepsis confirmed by positive blood culture
Necrotizing enterocolitis | first 28 days of life
  Necrotizing enterocolitis (Any Bell's stage)
Intraventricular hemorrhage | first 28 days of life
  Intraventricular hemorrhage of all grades
Bronchopulmonary dysplasia | first 70 days of life
  Oxygen requirement at 36 weeks corrected gestational age
Need for packed RBCs transfusion | first 28 days of life
  number of packed RBCs transfusion
Retinopathy of prematurity | first 28 days of life
  Prethreshold and threshold diseases Retinopathy of prematurity
Need for inotropes | first 28 days of life
  Hypotension requiring inotropic support
Need for nasal CPAP | first 28 days of life
  respiratory distress requiring CPAP support
Need for mechanical ventilation | first 28 days of life
  respiratory distress requiring mechanical ventilation support
Duration of oxygen therapy | first 70 days of life
  Duration of oxygen therapy

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura University Children Hospital, Al Mansurah, El Dakahlya
  - Mansoura University Children's Hospital, Al Mansurah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Yu B, Wang W, Luo D, Dai QL, Gan XQ. Does intact umbilical cord milking increase infection rates in preterm infants with premature prolonged rupture of membranes? J Matern Fetal Neonatal Med. 2020 Jan;33(2):184-190. doi: 10.1080/14767058.2018.1487947. Epub 2018 Sep 6. PMID 29886779
- [Result] Kumar B, Upadhyay A, Gothwal S, Jaiswal V, Joshi P, Dubey K. Umbilical Cord Milking and Hematological Parameters in Moderate to Late Preterm Neonates: A Randomized Controlled Trial. Indian Pediatr. 2015 Sep;52(9):753-7. doi: 10.1007/s13312-015-0711-1. PMID 26519708